CLINICAL TRIAL: NCT06559072
Title: Ultra-early STatin in Patients With Aneurysmal subaRachnoid Hemorrhage (Ue-STAR): a Randomized Controlled Trial
Brief Title: Ultra-early STatin in Patients With Aneurysmal subaRachnoid Hemorrhage (Ue-STAR)
Acronym: Ue-STAR
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: Tianjin Medical University General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2024-YX-167-01
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Subarachnoid Hemorrhage; Subarachnoid Hemorrhage, Aneurysmal; Aneurysmal Subarachnoid Hemorrhage; Hemorrhage, Aneurysmal Subarachnoid
Keywords: aneurysmal subarachnoid hemorrhage; atorvastatin; Atorvastatin Calcium
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Atorvastatin group (Experimental): On the basis of routine treatment for aneurysmal subarachnoid hemorrhage, atorvastatin was administered at an ultra early stage at a dose of 40mg/d for 14 consecutive days
  Interventions: Drug: Atorvastatin
- Conventional treatment group (No Intervention): Conventional treatment for aneurysmal subarachnoid hemorrhage typically includes measures such as blood pressure control, hemostasis, reduction of intracranial pressure, prevention of complications, and, when deemed necessary based on the patient's condition, surgical intervention. No specific interventions are applied unless warranted.

INTERVENTIONS:
Drug: Atorvastatin — On the basis of routine treatment for aneurysmal subarachnoid hemorrhage, atorvastatin was administered at an ultra early stage at a dose of 40mg/d for 14 consecutive days
  Arms: Atorvastatin group

SUMMARY:
A researcher-initiated and conducted multicenter, randomized controlled trial aimed at evaluating the efficacy and safety of ultra-early statin therapy in the treatment of acute aneurysmal subarachnoid hemorrhage (aSAH).

DETAILED DESCRIPTION:
To further explore the efficacy and safety of ultra-early statin administration in aSAH, the investigators propose a Phase III randomized controlled trial-The Ultra-early Statin in patients with Aneurysmal subArachnoid hemorrhage (Ue-STAR) trial. This study aims to determine whether ultra-early (within 6 hours), short-term treatment (2 weeks) with a high intensive long-acting statin (atorvastatin 40 mg/day) improves clinical outcomes at 6 months in aSAH patients. Through this research, the investigators hope to provide more robust evidence for the clinical management of aSAH, ultimately improving treatment outcomes for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; Aged ≥18 years
2. Signs and symptoms presumed aneurysmal subarachnoid hemorrhage, confirmed by radiological evidence
3. Treatment within 6 h after symptom onset

Exclusion Criteria:

1. Treatment with statin prior SAH
2. Non-aSAH (e.g. traumatic subarachnoid hemorrhage, arteriovenous malformation)
3. Treatment > 6 h after symptom onset
4. Allergy to statin medications or presence of severe adverse reactions such as abnormal liver function or rhabdomyolysis
5. Evidence of irreversible brain damage or expected death within 7 days
6. Known severe liver or kidney disease
7. Non-compliance with follow-up
8. Pregnant or breastfeeding
9. History of severe cranial or psychiatric illness
10. Concomitant serious systemic disease
11. Patients with malignant tumors
12. Currently participating in another clinical trial
13. Considered unsuitable for the clinical trial by clinical physicians or researchers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Utility-Weighted Modified Rankin Scale | 6 months after discharge
  A utility-weighted Modified Rankin Scale (UW-mRS) was derived by averaging values from time-tradeoff (patient centered) and person-tradeoff (clinician centered) studies. Utility values were 1.0 for Modified Rankin Scale (mRS) level 0; 0.91 for mRS level 1; 0.76 for mRS level 2; 0.65 for mRS level 3; 0.33 for mRS level 4; 0 for mRS level 5; and 0 for mRS level 6. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Modified Rankin Scale Score | 6 months after discharge
  The modified Rankin Scale (mRS) is the most widely used scale to measure the degree of handicap in stroke patients, ranging from 0 (no symptoms) to 6 (dead). Higher scores mean a worse outcome.
Glasgow Outcome Scale Extended | 6 months after discharge
  The Glasgow Outcome Scale Extended (GOS-E) is a clinical assessment tool used to assess outcome after head injury and nontraumatic acute brain insults. GOS-E divides patients' states into the following eight levels: dead, vegetative state, lower seven disability, upper seven disability, lower moderate disability, upper moderate disability, mild disability, lower good recovery, and basic recovery.
The 5-level EQ-5D version | 6 months after discharge
  The 5-level EQ-5D version (EQ-5D-5L) essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled "The best health you can image" and "The worst health you can image".

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes
After a domain is completed, the archived de-identified limited dataset of randomized participants will be transmitted to and stored in the Data Repository, for use by researchers. Data can be shared after publication of the main results unless specified otherwise in domain-specific registration.
Supporting Information: Study Protocol
Time Frame: Open data access within 12 months after the publication of research results
Access Criteria: Data can be shared after publication of the main results, based on approval of a submitted protocol to the Publication Committee. Data can be shared to bona fide researchers with experience in medical research, and with no conflict of interest that may potentially influence their interpretation of any analyses, and employed by a recognised academic institute, health service organisation, commercial research organisation of from the pharmaceutical industry. The data sharing will be only for analyses within the constraints of the consent under which the data were originally gathered consent.
  Data sharing with industry will be according to relevant contracts with appropriate approvals from all stake holders.
URL: https://dct-dev.meddb.cn